CLINICAL TRIAL: NCT01854632
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of the Clinical Efficacy of Trivalent Live-Attenuated Influenza Vaccine (LAIV) Among Children in Senegal
Brief Title: Clinical Efficacy of Trivalent Live-Attenuated Influenza Vaccine (LAIV) Among Children in Senegal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Institut de Recherche pour le Developpement (Other Government); Institut Pasteur de Dakar (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAIV-SEN-01
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-02

CONDITIONS: Influenza
Keywords: influenza vaccine; trivalent live-attenuated influenza vaccine; efficacy; Africa; Senegal
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIIL Live Attenuated Influenza Vaccine (Experimental): Single 0.5 mL dose of trivalent live-attenuated influenza vaccine 2012/2013 Northern Hemisphere vaccine containing A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010
  Interventions: Biological: SIIL Live Attenuated Influenza Vaccine
- Matched placebo (Placebo Comparator): Single 0.5mL inactive placebo will be identical to reconstituted SIIL LAIV in ingredients and concentrations except A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010 will be replaced with egg allantoic fluid.
  Interventions: Biological: Matched placebo

INTERVENTIONS:
Biological: SIIL Live Attenuated Influenza Vaccine — Trivalent live-attenuated influenza vaccine 2012/2013 Northern Hemisphere vaccine containing A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010
  Arms: SIIL Live Attenuated Influenza Vaccine
Biological: Matched placebo — Matched placebo will be identical to reconstituted SIIL LAIV in ingredients and concentrations except A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010 will be replaced with egg allantoic fluid.
  Arms: Matched placebo

SUMMARY:
This study will provide the Senegal Ministry of Health with data on the clinical efficacy of the Live-Attenuated Influenza Vaccine (LAIV). This data will inform future policy considerations for influenza vaccine.

DETAILED DESCRIPTION:
This study is a double-blind, individual-randomized, placebo-controlled, clinical efficacy trial among healthy children aged 24 through 71 months in the Niakhar area of Senegal. A total of 1,761 healthy children will be randomized in a 2:1 ratio of LAIV to placebo.

For evaluation of efficacy, passive and active surveillance will be conducted weekly throughout the study to identify outcomes among vaccinated subjects. Children meeting the protocol-defined clinical case definition will have a nasal swab and throat swab specimen collected for testing by rRT-PCR for evidence of influenza virus infection.

100 of the 1,761 participants were also included in a substudy designed to evaluate virologic evidence of LAIV replication. As such, nasal and throat swab specimens were collected on day 0 (prior to vaccination), as well as on post-vaccination days 2, and 4 from all subjects included in the substudy. These specimens will be tested for presence of wild-type and vaccine virus. Additionally, a more detailed assessment of vaccine reactogenicity will be made among these children by actively collecting solicited and unsolicited reactions at each study visit for the week post vaccination (days 2 and 4).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female child at least 24 months of age and no older than 71 months of age at the time of study vaccination.
* A child whose parent or guardian's primary residence, at the time of study vaccinations, is within the Niakhar DSS and who intends to be present in the area for the duration of the trial.
* A child whose parent or legal guardian is willing to provide written informed consent prior to the participant's study vaccination

Exclusion Criteria:

* Serious, active, medical condition, including: chronic disease of any body system,chronic infections such as tuberculosis, genetic disorders, such as Down's syndrome or other cytogenetic disorder, known or suspected disease of the immune system of any kind.
* History of documented hypersensitivity to eggs or other components of the vaccine (including gelatin, sorbitol, lactalbumin and chicken protein), or with life-threatening reactions to previous influenza vaccinations.
* History of Guillain-Barré syndrome.
* Receipt of immunosuppressive agents, including systemic corticosteroids, during the month before planned study vaccination.
* Receipt of aspirin therapy or aspirin-containing therapy within the two weeks before planned study vaccination.
* History of any severe allergic reaction with generalized urticarial, angioedema, or anaphylaxis.
* Receipt of an influenza vaccine within the past 12 months.
* Has any condition determined by investigator as likely to interfere with evaluation of the vaccine or be a significant potential health risk to the child or make it unlikely that the child would complete the study.

Temporary Contraindications:

* Acute illness accompanied by a body temperature of 37.5°C or above (axillary measurement) within 14 days of enrollment visit.
* Any acute respiratory infection within 14 days of enrollment visit.
* Any illness accompanied by active wheezing within 14 days of enrollment visit.

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1761 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aldiouma Diallo, MD, Principal Investigator — Institut de Recherche pour le Développement (IRD)
Locations (1):
- Institut de Recherche pour le Développement (IRD), Niakhar station, Niakhar, Senegal

REFERENCES:
- [Derived] Victor JC, Lewis KD, Diallo A, Niang MN, Diarra B, Dia N, Ortiz JR, Widdowson MA, Feser J, Hoagland R, Emery SL, Lafond KE, Neuzil KM. Efficacy of a Russian-backbone live attenuated influenza vaccine among children in Senegal: a randomised, double-blind, placebo-controlled trial. Lancet Glob Health. 2016 Dec;4(12):e955-e965. doi: 10.1016/S2214-109X(16)30201-7. Epub 2016 Oct 13. PMID 27746224

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine: Single dose of trivalent live-attenuated influenza vaccine 2012/2013 Northern Hemisphere vaccine containing A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010
- Placebo: Single dose of placebo will be identical to reconstituted SIIL LAIV in ingredients and concentrations except A/California/7/2009 (H1N1), A/Victoria/361/2011 (H3N2), B/Wisconsin/1/2010 will be replaced with egg allantoic fluid.
Period: Overall Study
Arm/Group | Vaccine | Placebo
Started | 1174 | 587
Completed | 1148 | 574
Not Completed | 26 | 13

BASELINE CHARACTERISTICS:
Population: All enrolled participants receiving the single dose of study vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 1174 | 587 | 1761
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1174 | 587 | 1761
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 564 | 290 | 854
  Male | 610 | 297 | 907
Region of Enrollment [Number; unit: participants]
  Senegal | 1174 | 587 | 1761

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed Influenza Virus Infection (Regardless of Vaccine Match)
Time Frame: Through 7 to 8 months post vaccination
Population: All participants meeting per-protocol analysis criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1173 | 584
percentage of participants | 17.9 | 18.0
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Superiority or Other; p = 0.996, Log Rank

2. Secondary Outcome: Safety Profile of LAIV: Immediate Reactions Occurring Within 30 Minutes of Administration of Study Vaccine.
Time Frame: Through 30 minutes post vaccination
Reporting Status: Not Posted

3. Secondary Outcome: Safety Profile of LAIV: Solicited and Unsolicited Local and Systemic Reactions
Time Frame: Through 7 days post vaccination
Reporting Status: Not Posted

4. Secondary Outcome: Safety Profile of LAIV: Serious Adverse Events
Time Frame: Through 1 month post vaccination
Reporting Status: Not Posted

5. Secondary Outcome: Safety Profile of LAIV: Other Non-serious Adverse Events
Time Frame: Through 1 month post vaccination
Reporting Status: Not Posted

6. Secondary Outcome: Safety Profile of LAIV: Protocol Defined Wheezing Illness
Time Frame: Through 7 to 8 months post vaccination
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed Influenza Virus Infection (Vaccine-matched Strains)
Time Frame: Through 7 to 8 months post vaccination
Reporting Status: Not Posted

8. Secondary Outcome: Percentage of Participants With Symptomatic, Laboratory-confirmed Influenza Virus Infection by Influenza Type/Subtype (Influenza A/H1N1, Influenza A/H3N2, and Influenza B)
Time Frame: Through 7 to 8 months post vaccination
Reporting Status: Not Posted

9. Secondary Outcome: Clinical Characteristics of Influenza in the Study Population
Time Frame: Through 7 to 8 months post vaccination
Reporting Status: Not Posted

10. Secondary Outcome: Etiologies of Influenza-like Illness in the Study Population
Description: Bacterial and viral etiologies of acute respiratory and febrile illness will be parameterized as the percentage of those with each particular laboratory-confirmed infection categorized by vaccine allocation.
Time Frame: Through 7 to 8 months post vaccination
Reporting Status: Not Posted

11. Secondary Outcome: Evaluation of Vaccine-take as Shedding of Vaccine Virus Post-vaccination, Including Viral Load and Duration of Virus Detection
Description: Vaccine take will be parameterized as the percentage of participants with detectable vaccine-virus in nasal or throat swab on each day pre- (day 0) and post vaccination (i.e., 2 and 4 days post vaccination), and the quantity of detected virus.
Time Frame: Through 4 days post vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout the study period: May through December 2013
Arm/Group | Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 7/1174 | 7/587
Other Adverse Events (participants affected / at risk) | 56/1174 | 33/587
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=1174) | Placebo (N=587)
Trauma (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Respiratory illnesses (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Other (General disorders) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=1174) | Placebo (N=587)
Respiratory AEs (Respiratory, thoracic and mediastinal disorders) | 17 | 16
Non Respiratory AEs (General disorders) | 39 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less